CLINICAL TRIAL: NCT03080103
Title: A Prospective Non-randomized Controlled, Multicenter, Multidisciplinary Trial Comparing Appendectomy and Conservative Treatment for Patients With Uncomplicated Acute Appendicitis (the ACTUAA STUDY).
Brief Title: Appendectomy Versus Conservative Treatment for Uncomplicated Acute Appendicitis
Acronym: ACTUAA
Status: Completed | Type: Observational
Sponsor: Mauro Podda (Other)
Collaborators: Associazione Chirurghi Ospedalieri Italiani (Other)
Responsible Party: Sponsor-Investigator, Mauro Podda, Dr. Mauro Podda, M.D., Associazione Chirurghi Ospedalieri Italiani
Organization: Associazione Chirurghi Ospedalieri Italiani (Other)
Other Study IDs: No ID
Record Dates: First submitted 2017-03-05; First posted 2017-03-15 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Acute Appendicitis; Appendicitis Recurrent; Appendectomy; Antibiotic Therapy
Keywords: Acute Appendicitis; Uncomplicated Acute Appendicitis; Appendectomy; Conservative Treatment; Antibiotic-first Treatment; Recurrent Appendicitis; Prospective Study
MeSH Terms: conditions — Appendicitis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens of the appendix
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients submitted to appendectomy as first-line treatment: Open or Laparoscopic Appendectomy The assignment of each patient to either the "antibiotic-first management" arm or the "immediate surgery" arm, will be non-randomized and decided independently by the Staff Specialist Surgeon on Call, upon careful assessment of AIR score, laboratory findings and imaging. The decision of the management pathway will not be influenced in any case by the participation of the patient in the study, and the assignment of the treatment will be decided by the consultant surgeon according to current good surgical practice and standard practice patterns in Italy.
  Interventions: Procedure: Laparoscopic or Open appendectomy
- Patients treated with antibiotic-first strategy: Antibiotic therapy.maging. Patients managed conservatively will receive one of the following parenteral antibiotic treatments: Piperacillin/Tazobactam (4.5 g) three intravenous administration per day; Ceftriaxone (2 g) once per day or Ciprofloxacin (500 mg) twice per day plus Metronidazole (500 mg) three times per day; Amoxicillin/Clavulanic acid (2 g) four times per day for a length depending on the clinical conditions; Ertapenem (1 g) one administration per day for three days. Patients were discharged with oral antibiotics (amoxicillin/clavulanic acid or ciprofloxacin) for at least four days.
  Interventions: Drug: Antibiotic-first therapy

INTERVENTIONS:
Procedure: Laparoscopic or Open appendectomy — Laparoscopic three-port or single-port appendectomy; or conventional McBurney laparotomic appendectomy; or open appendectomy performed through midline incision
  Groups: Patients submitted to appendectomy as first-line treatment
Drug: Antibiotic-first therapy — Patients treated with antibiotics as first-line approach
  Groups: Patients treated with antibiotic-first strategy

SUMMARY:
On September the 15th, 2015, Italian surgeons, radiologists and pathologists with a special interest and expertise in the diagnosis and management of Acute Appendicitis (AA), met up under the auspices of the Italian Society of Hospital Surgeons (ACOI) in Oristano (Italy) to constitute the ACTUAA collaborative working group. The main objectives of the working group are:

To create a working basis for analyzing the diagnostic features, treatment modalities and outcomes of interest of both the antibiotic-first approach and appendectomy for patients with uncomplicated AA.

To investigate the clinical, laboratory and radiologic modalities adopted for the diagnosis To determine the outcomes of patients treated with antibiotics or appendectomy in the short and long term periods.

To compare results according to the type of intervention. To stratify the risk of recurrence for patients treated with antibiotics according to clinical, laboratory and radiology findings.

To evaluate the sensibility and specificity of clinical and laboratory scores for the diagnosis of uncomplicated AA.

To identify a subgroup of patients with uncomplicated AA for whom antibiotic treatment can be highly effective.

General study design The study protocol is designed according to the "SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials".

The study period is estimated to be of 12 month + 12 month of follow-up (with a second session of follow-up following 5-years), beginning on 01/04/2017.

Participants All adult patients (aged over 18 years old) with suspected AA will be admitted to the Surgical Department of the nine participating Italian hospitals, where they will be studied carefully by the on call surgeon.

Patients will be then informed of the study protocol and invited to give written consent for participation and for sensible data collection for scientific purposes.

Subsequently, only patients who will undergo diagnostic imaging (as specified later) and from whom a written informed consent will be obtained, can be enrolled in the study and registered by each Center using a uniform electronic registration form and database.

General characteristics, medical history, clinical findings, physical investigation, and blood tests will be reported in the medical record. Pain will be quantified by Visual Analogue Scale (VAS) scoring system before administrating any pain medications and after the treatments.

In order to enter the study, patients will have to undergo diagnostic imaging (US and/or CT scan or MRI scan) and only the diagnosis of uncomplicated AA confirmed by diagnostic imaging will permit patient enrollment in the study.

Specific aims of the ACTUAA Study The objective of this prospective non-randomized controlled, multicenter, multidisciplinary trial is to compare the antibiotic therapy and emergency appendectomy for the treatment of patients with uncomplicated AA(without abscess or free perforation), confirmed by US and/or CT or MRI scan. No changes in the daily practice regarding the diagnostic, clinical and treatment pathways will be required to the participating centers. However, only the patients with uncomplicated AA, confirmed by one of the above mentioned radiologic tools will be enrolled in the study. The decision on which of the tools are to be adopted will be up to the local lead surgeon.

Primary Outcome Measure:

Number of participants with complication-free treatment success, defined as success of the initial treatment with uncomplicated course.

Secondary Outcome Measures:

Length of hospital stay; Pain evaluation; Time to return to normal activity; Period of sick-leave; Complicated appendicitis with peritonitis identified at the time of surgical operation; Quality of life as assessed by the Short Form 12-scale (SF-12)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age over 18 years
* Uncomplicated AA confirmed by US and/or CT or MRI scan.

Exclusion Criteria:

* Pregnancy or lactating
* Diffuse peritonitis at physical examination
* Serious systemic illness
* Positive anamnesis for Inflammatory Bowel Disease (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (aged over 18 years old) with suspected Acute Appendicitis admitted to the Surgical Department of the nine participating Italian Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with complication-free treatment success, as assessed by the Dindo-Clavien Scale. | 1 year
  Number of participants with complication-free treatment success, defined as success of the initial treatment with uncomplicated course: no postoperative complications, adverse events, or treatment failure occurring, as assessed by the Dindo-Clavien Classification. Post-treatment abdominal abscess, bowel occlusion, incisional hernia, pulmonary embolism, cardio-vascular complications, surgical site infection, complications due to anesthesia, adverse reactions to antibiotics. Complications are analyzed both for patients submitted to appendectomy and for those treated with surgery as second line approach, after primary antibiotic treatment failure. For patients treated with antibiotics, treatment failure (persistency and recurrence rates of acute appendicitis) will be evaluated within the overall-complications rate. Specific sub-analyses of the complications will be carried out.

SECONDARY OUTCOMES:
Length of hospital stay | 1 week
  Length of post-operative hospital stay for patients submitted to appendectomy; length of hospital stay for patients treated with antibiotics
VAS-Score | 1 month
  Pain evaluation performed through the visual analogue scale both for patients who undergo an appendectomy and for those treated with antibiotics
Time to return to normal activity | 1 month
  Time to return to normal activity both for patients who undergo an appendectomy and for those treated with antibiotics
Period of sick-leave | 1 month
  Period of sick-leave, intended as "absence from work"
Complicated appendicitis with peritonitis identified at the time of surgical operation. | 1 year
  In the antibiotic group the analysis will be carried out within the cohort of patients who will undergo appendectomy after the failure of the antibiotic therapy in order to assess whether or not a major risk of perforated appendicitis exists for patients who will be treated firstly with antibiotics.
Quality of life as assessed by the Short Form 12-scale (SF-12) | 1 year
  Quality of life estimated by the Short Form 12-scale (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Podda, M.D., Study Director — Associazione dei Chirurghi Ospedalieri Italiani ACOI; General Surgeon, San Francesco Hospital. Nuoro (Italy)
Locations (7):
- Italy (7):
  - General and Emergency Surgery Unit, San Marcellino Hospital, Muravera, Cagliari
  - Department of General Surgery, San Giovanni Addolorata Hospital, Rome, Italt
  - General Surgery Unit, Nostra Signora Della Mercede Hospita, Lanusei, Lanusei, Ogliastra
  - General and Endocrine Surgical Unit, Cagliari University Hospital, Cagliari, Cagliari
  - General Surgery, Santissima Trinità Hospital, Cagliari
  - Emergency Surgery Unit, Villa Betania Evangelic Hospital, Napoli, Napoli
  - General, Minimally Invasive and Robotic Surgery, San Francesco Hospital, Nuoro

IPD SHARING:
Plan to Share IPD: No
Data will be published as a pool from all participating surgical units. Subgroup analysis by grade of the disease based on the AIR score, surgical technique, histological grade of the appendicitis, type of antibiotic used or outcome variables may be presented, but, in order to avoid the identification of an individual unit or surgeon, no hospital level or surgeon level data will be published.Each participating centre, with equal right, will be able to access the data of the registry, perform statistical analysis, discuss the results and freely write scientific manuscripts. Each study that is generated based on the registry must be disseminated to all the centres before final publication.

REFERENCES:
- [Background] DeFrances CJ, Hall MJ. 2002 National Hospital Discharge Survey. Adv Data. 2004 May 21;(342):1-29. PMID 15174387
- [Background] Livingston EH, Woodward WA, Sarosi GA, Haley RW. Disconnect between incidence of nonperforated and perforated appendicitis: implications for pathophysiology and management. Ann Surg. 2007 Jun;245(6):886-92. doi: 10.1097/01.sla.0000256391.05233.aa. PMID 17522514
- [Background] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906
- [Background] Di Saverio S, Birindelli A, Kelly MD, Catena F, Weber DG, Sartelli M, Sugrue M, De Moya M, Gomes CA, Bhangu A, Agresta F, Moore EE, Soreide K, Griffiths E, De Castro S, Kashuk J, Kluger Y, Leppaniemi A, Ansaloni L, Andersson M, Coccolini F, Coimbra R, Gurusamy KS, Campanile FC, Biffl W, Chiara O, Moore F, Peitzman AB, Fraga GP, Costa D, Maier RV, Rizoli S, Balogh ZJ, Bendinelli C, Cirocchi R, Tonini V, Piccinini A, Tugnoli G, Jovine E, Persiani R, Biondi A, Scalea T, Stahel P, Ivatury R, Velmahos G, Andersson R. WSES Jerusalem guidelines for diagnosis and treatment of acute appendicitis. World J Emerg Surg. 2016 Jul 18;11:34. doi: 10.1186/s13017-016-0090-5. eCollection 2016. PMID 27437029
- [Background] Agresta F, Campanile FC, Podda M, Cillara N, Pernazza G, Giaccaglia V, Ciccoritti L, Ioia G, Mandala S, La Barbera C, Birindelli A, Sartelli M, Di Saverio S; Joined Italian Surgical Societies Working Group. Current status of laparoscopy for acute abdomen in Italy: a critical appraisal of 2012 clinical guidelines from two consecutive nationwide surveys with analysis of 271,323 cases over 5 years. Surg Endosc. 2017 Apr;31(4):1785-1795. doi: 10.1007/s00464-016-5175-4. Epub 2016 Aug 29. PMID 27572068
- [Background] Sartelli M, Catena F, Ansaloni L, Coccolini F, Griffiths EA, Abu-Zidan FM, Di Saverio S, Ulrych J, Kluger Y, Ben-Ishay O, Moore FA, Ivatury RR, Coimbra R, Peitzman AB, Leppaniemi A, Fraga GP, Maier RV, Chiara O, Kashuk J, Sakakushev B, Weber DG, Latifi R, Biffl W, Bala M, Karamarkovic A, Inaba K, Ordonez CA, Hecker A, Augustin G, Demetrashvili Z, Melo RB, Marwah S, Zachariah SK, Shelat VG, McFarlane M, Rems M, Gomes CA, Faro MP, Junior GA, Negoi I, Cui Y, Sato N, Vereczkei A, Bellanova G, Birindelli A, Di Carlo I, Kok KY, Gachabayov M, Gkiokas G, Bouliaris K, Colak E, Isik A, Rios-Cruz D, Soto R, Moore EE. WSES Guidelines for the management of acute left sided colonic diverticulitis in the emergency setting. World J Emerg Surg. 2016 Jul 29;11:37. doi: 10.1186/s13017-016-0095-0. eCollection 2016. PMID 27478494
- [Background] Katkhouda N, Mason RJ, Towfigh S, Gevorgyan A, Essani R. Laparoscopic versus open appendectomy: a prospective randomized double-blind study. Ann Surg. 2005 Sep;242(3):439-48; discussion 448-50. doi: 10.1097/01.sla.0000179648.75373.2f. PMID 16135930
- [Background] Di Saverio S, Sartelli M, Catena F, Birindelli A, Tugnoli G. Renewed Interest in Acute Appendicitis: Are Antibiotics Non-Inferior to Surgery or Possibly Clinically Superior? What Is Long-Term Follow-Up and Natural Evolution of Appendicitis Treated Conservatively with "Antibiotics First"? Surg Infect (Larchmt). 2016 Jun;17(3):376-7. doi: 10.1089/sur.2015.206. Epub 2016 Feb 26. No abstract available. PMID 26918798
- [Background] Liu K, Fogg L. Use of antibiotics alone for treatment of uncomplicated acute appendicitis: a systematic review and meta-analysis. Surgery. 2011 Oct;150(4):673-83. doi: 10.1016/j.surg.2011.08.018. PMID 22000179
- [Background] Nakhamiyayev V, Galldin L, Chiarello M, Lumba A, Gorecki PJ. Laparoscopic appendectomy is the preferred approach for appendicitis: a retrospective review of two practice patterns. Surg Endosc. 2010 Apr;24(4):859-64. doi: 10.1007/s00464-009-0678-x. PMID 19730948
- [Background] Flum DR, Koepsell T. The clinical and economic correlates of misdiagnosed appendicitis: nationwide analysis. Arch Surg. 2002 Jul;137(7):799-804; discussion 804. doi: 10.1001/archsurg.137.7.799. PMID 12093335
- [Background] Styrud J, Eriksson S, Nilsson I, Ahlberg G, Haapaniemi S, Neovius G, Rex L, Badume I, Granstrom L. Appendectomy versus antibiotic treatment in acute appendicitis. a prospective multicenter randomized controlled trial. World J Surg. 2006 Jun;30(6):1033-7. doi: 10.1007/s00268-005-0304-6. PMID 16736333
- [Background] Turhan AN, Kapan S, Kutukcu E, Yigitbas H, Hatipoglu S, Aygun E. Comparison of operative and non operative management of acute appendicitis. Ulus Travma Acil Cerrahi Derg. 2009 Sep;15(5):459-62. PMID 19779986
- [Background] Vons C, Barry C, Maitre S, Pautrat K, Leconte M, Costaglioli B, Karoui M, Alves A, Dousset B, Valleur P, Falissard B, Franco D. Amoxicillin plus clavulanic acid versus appendicectomy for treatment of acute uncomplicated appendicitis: an open-label, non-inferiority, randomised controlled trial. Lancet. 2011 May 7;377(9777):1573-9. doi: 10.1016/S0140-6736(11)60410-8. PMID 21550483
- [Background] Podda M, Cillara N, Di Saverio S, Lai A, Feroci F, Luridiana G, Agresta F, Vettoretto N; ACOI (Italian Society of Hospital Surgeons) Study Group on Acute Appendicitis. Antibiotics-first strategy for uncomplicated acute appendicitis in adults is associated with increased rates of peritonitis at surgery. A systematic review with meta-analysis of randomized controlled trials comparing appendectomy and non-operative management with antibiotics. Surgeon. 2017 Oct;15(5):303-314. doi: 10.1016/j.surge.2017.02.001. Epub 2017 Mar 9. PMID 28284517
- [Background] Wilms IM, de Hoog DE, de Visser DC, Janzing HM. Appendectomy versus antibiotic treatment for acute appendicitis. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD008359. doi: 10.1002/14651858.CD008359.pub2. PMID 22071846
- [Background] Findlay JM, Kafsi JE, Hammer C, Gilmour J, Gillies RS, Maynard ND. Nonoperative Management of Appendicitis in Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Coll Surg. 2016 Dec;223(6):814-824.e2. doi: 10.1016/j.jamcollsurg.2016.09.005. Epub 2016 Oct 26. No abstract available. PMID 27793458
- [Background] Salminen P, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Tuominen R, Hurme S, Virtanen J, Mecklin JP, Sand J, Jartti A, Rinta-Kiikka I, Gronroos JM. Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis: The APPAC Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2340-8. doi: 10.1001/jama.2015.6154. PMID 26080338
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Harnoss JC, Zelienka I, Probst P, Grummich K, Muller-Lantzsch C, Harnoss JM, Ulrich A, Buchler MW, Diener MK. Antibiotics Versus Surgical Therapy for Uncomplicated Appendicitis: Systematic Review and Meta-analysis of Controlled Trials (PROSPERO 2015: CRD42015016882). Ann Surg. 2017 May;265(5):889-900. doi: 10.1097/SLA.0000000000002039. PMID 27759621
- [Background] Andersson M, Andersson RE. The appendicitis inflammatory response score: a tool for the diagnosis of acute appendicitis that outperforms the Alvarado score. World J Surg. 2008 Aug;32(8):1843-9. doi: 10.1007/s00268-008-9649-y. PMID 18553045
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Eriksson S, Granstrom L. Randomized controlled trial of appendicectomy versus antibiotic therapy for acute appendicitis. Br J Surg. 1995 Feb;82(2):166-9. doi: 10.1002/bjs.1800820207. PMID 7749676
- [Background] Hansson J, Korner U, Khorram-Manesh A, Solberg A, Lundholm K. Randomized clinical trial of antibiotic therapy versus appendicectomy as primary treatment of acute appendicitis in unselected patients. Br J Surg. 2009 May;96(5):473-81. doi: 10.1002/bjs.6482. PMID 19358184
- [Background] Gregory S, Kuntz K, Sainfort F, Kharbanda A. Cost-Effectiveness of Integrating a Clinical Decision Rule and Staged Imaging Protocol for Diagnosis of Appendicitis. Value Health. 2016 Jan;19(1):28-35. doi: 10.1016/j.jval.2015.10.007. Epub 2015 Dec 2. PMID 26797233
- [Background] Sammalkorpi HE, Mentula P, Leppaniemi A. A new adult appendicitis score improves diagnostic accuracy of acute appendicitis--a prospective study. BMC Gastroenterol. 2014 Jun 26;14:114. doi: 10.1186/1471-230X-14-114. PMID 24970111
- [Background] Rao PM, Rhea JT, Novelline RA, Mostafavi AA, McCabe CJ. Effect of computed tomography of the appendix on treatment of patients and use of hospital resources. N Engl J Med. 1998 Jan 15;338(3):141-6. doi: 10.1056/NEJM199801153380301. PMID 9428814
- [Background] van Randen A, Lameris W, van Es HW, van Heesewijk HP, van Ramshorst B, Ten Hove W, Bouma WH, van Leeuwen MS, van Keulen EM, Bossuyt PM, Stoker J, Boermeester MA; OPTIMA Study Group. A comparison of the accuracy of ultrasound and computed tomography in common diagnoses causing acute abdominal pain. Eur Radiol. 2011 Jul;21(7):1535-45. doi: 10.1007/s00330-011-2087-5. Epub 2011 Mar 2. PMID 21365197
- [Background] Humes DJ, Simpson J. Acute appendicitis. BMJ. 2006 Sep 9;333(7567):530-4. doi: 10.1136/bmj.38940.664363.AE. No abstract available. PMID 16960208
- [Background] Jones RP, Jeffrey RB, Shah BR, Desser TS, Rosenberg J, Olcott EW. Journal Club: the Alvarado score as a method for reducing the number of CT studies when appendiceal ultrasound fails to visualize the appendix in adults. AJR Am J Roentgenol. 2015 Mar;204(3):519-26. doi: 10.2214/AJR.14.12864. PMID 25714280
- [Background] Lameris W, van Randen A, van Es HW, van Heesewijk JP, van Ramshorst B, Bouma WH, ten Hove W, van Leeuwen MS, van Keulen EM, Dijkgraaf MG, Bossuyt PM, Boermeester MA, Stoker J; OPTIMA study group. Imaging strategies for detection of urgent conditions in patients with acute abdominal pain: diagnostic accuracy study. BMJ. 2009 Jun 26;338:b2431. doi: 10.1136/bmj.b2431. PMID 19561056
- [Background] Krishnamoorthi R, Ramarajan N, Wang NE, Newman B, Rubesova E, Mueller CM, Barth RA. Effectiveness of a staged US and CT protocol for the diagnosis of pediatric appendicitis: reducing radiation exposure in the age of ALARA. Radiology. 2011 Apr;259(1):231-9. doi: 10.1148/radiol.10100984. Epub 2011 Jan 28. PMID 21324843
- [Background] Nielsen JW, Boomer L, Kurtovic K, Lee E, Kupzyk K, Mallory R, Adler B, Bates DG, Kenney B. Reducing computed tomography scans for appendicitis by introduction of a standardized and validated ultrasonography report template. J Pediatr Surg. 2015 Jan;50(1):144-8. doi: 10.1016/j.jpedsurg.2014.10.033. Epub 2014 Dec 18. PMID 25598112
- [Background] Aspelund G, Fingeret A, Gross E, Kessler D, Keung C, Thirumoorthi A, Oh PS, Behr G, Chen S, Lampl B, Middlesworth W, Kandel J, Ruzal-Shapiro C. Ultrasonography/MRI versus CT for diagnosing appendicitis. Pediatrics. 2014 Apr;133(4):586-93. doi: 10.1542/peds.2013-2128. Epub 2014 Mar 3. PMID 24590746
- [Background] Rettenbacher T, Hollerweger A, Macheiner P, Rettenbacher L, Frass R, Schneider B, Gritzmann N. Presence or absence of gas in the appendix: additional criteria to rule out or confirm acute appendicitis--evaluation with US. Radiology. 2000 Jan;214(1):183-7. doi: 10.1148/radiology.214.1.r00ja20183. PMID 10644120
- [Background] Mostbeck G, Adam EJ, Nielsen MB, Claudon M, Clevert D, Nicolau C, Nyhsen C, Owens CM. How to diagnose acute appendicitis: ultrasound first. Insights Imaging. 2016 Apr;7(2):255-63. doi: 10.1007/s13244-016-0469-6. Epub 2016 Feb 16. PMID 26883138
- [Background] Quigley AJ, Stafrace S. Ultrasound assessment of acute appendicitis in paediatric patients: methodology and pictorial overview of findings seen. Insights Imaging. 2013 Dec;4(6):741-51. doi: 10.1007/s13244-013-0275-3. Epub 2013 Aug 31. PMID 23996381
- [Background] Birnbaum BA, Wilson SR. Appendicitis at the millennium. Radiology. 2000 May;215(2):337-48. doi: 10.1148/radiology.215.2.r00ma24337. PMID 10796905
- [Background] Incesu L, Yazicioglu AK, Selcuk MB, Ozen N. Contrast-enhanced power Doppler US in the diagnosis of acute appendicitis. Eur J Radiol. 2004 May;50(2):201-9. doi: 10.1016/S0720-048X(03)00102-5. PMID 15081132
- [Background] Shogilev DJ, Duus N, Odom SR, Shapiro NI. Diagnosing appendicitis: evidence-based review of the diagnostic approach in 2014. West J Emerg Med. 2014 Nov;15(7):859-71. doi: 10.5811/westjem.2014.9.21568. Epub 2014 Oct 7. PMID 25493136
- [Background] Karul M, Berliner C, Keller S, Tsui TY, Yamamura J. Imaging of appendicitis in adults. Rofo. 2014 Jun;186(6):551-8. doi: 10.1055/s-0034-1366074. Epub 2014 Apr 23. PMID 24760428
- [Background] Bixby SD, Lucey BC, Soto JA, Theysohn JM, Ozonoff A, Varghese JC. Perforated versus nonperforated acute appendicitis: accuracy of multidetector CT detection. Radiology. 2006 Dec;241(3):780-6. doi: 10.1148/radiol.2413051896. PMID 17114626
- [Background] Ramdass MJ, Young Sing Q, Milne D, Mooteeram J, Barrow S. Association between the appendix and the fecalith in adults. Can J Surg. 2015 Feb;58(1):10-4. doi: 10.1503/cjs.002014. PMID 25427333
- [Derived] Podda M, Poillucci G, Pacella D, Mortola L, Canfora A, Aresu S, Pisano M, Erdas E, Pisanu A, Cillara N; ACTUAA Study Collaborative Working Group. Appendectomy versus conservative treatment with antibiotics for patients with uncomplicated acute appendicitis: a propensity score-matched analysis of patient-centered outcomes (the ACTUAA prospective multicenter trial). Int J Colorectal Dis. 2021 Mar;36(3):589-598. doi: 10.1007/s00384-021-03843-8. Epub 2021 Jan 17. PMID 33454817
- [Derived] Podda M, Serventi F, Mortola L, Marini S, Sirigu D, Piga M, Pisano M, Coppola M, Agresta F, Virdis F, Di Saverio S, Cillara N; ACTUAA Study Collaborative Working Group. A prospective non-randomized controlled, multicenter trial comparing Appendectomy and Conservative Treatment for Patients with Uncomplicated Acute Appendicitis (the ACTUAA study). Int J Colorectal Dis. 2017 Nov;32(11):1649-1660. doi: 10.1007/s00384-017-2878-5. Epub 2017 Aug 15. PMID 28812175